CLINICAL TRIAL: NCT06999551
Title: Comparison of the Efficacy and Safety of GLARGEN® Versus NPH Insulin in the Treatment of Diabetes Type 2, in Tunisian Patients.
Brief Title: Comparison of the Efficacy and Safety of GLARGEN® Versus NPH Insulin in Diabetic Tunisian Patients.
Acronym: GRANT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRANT2025
Record Dates: First submitted 2025-03-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; NPH; Insulin glargin; continuous glucose monitoring; efficacy; safety
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient receiving NPH insulin (Experimental): evaluating safety and efficacy after switching the patient receiving NPH into glargin insulin.
  Interventions: Drug: switch NPH to glargin

INTERVENTIONS:
Drug: switch NPH to glargin — Switch of patients with type 2 diabetes mellitus from NPH insulin to insulin glargine

SUMMARY:
This study will have a single arm: the patient on NPH will continue his treatment for 4 weeks, at the end of the NPH treatment, the patient will receive his CGM device for three days for glycemic holter, a switch to insulin glargine is started for a period of 12 weeks with a dose adjustment and a control of the glycemic balance by CGM for three days at the end of the study.

The NPH insulin vial is a 10 ml vial dosed at 100 IU/mL, The Glargen vial is in the form of a solution for injection, a 3 ml vial dosed at 100 IU/mL

DETAILED DESCRIPTION:
Follow-up visits will include :

* V0: - 4 weeks: Screening visit (before the start of treatment): patients will be selected at this initial visit, if they meet all the inclusion criteria and none of the non-inclusion criteria, the patient will receive the glucometer. The patient presents himself to do his initial assessment (including HbA1c) and sign the consent, to do his therapeutic education and to receive the nutrition booklet
* V1: -3 weeks: the patient will be contacted by the ARC (phone call) to communicate the results of the glycemic cycle already performed and for titration of his NPH, continue with the new dose until the monitoring stops
* V2: inclusion visit: D0: 4 weeks later, the patient will receive his CGM. A glycemic cycle will be done and communicated to the ARC.
* V3: Visit of 4 weeks + 07 days: the day the patient presents himself to put the CGM device back on (stop monitoring) and collect data (glycemic holter under NPH) and switch to insulin glargine.
* V4 + V5: respectively at 2 and 3 weeks after switching to insulin glargine, the CRA contacts the patient by phone to record the results of the glycemic cycle and thus adapt the dose of insulin glargine upwards or downwards as needed (titration). The patient will do a glycemic cycle and communicate it to their ARC. Continue with the new dose until the next V6 titration
* V6: at 6 weeks after switching to insulin glargine, the patient will attend the consultation (face-to-face) to communicate the results of the corresponding glycemic cycle and thus adapt the dose of insulin glargine upwards or downwards as needed (titration). Continue with the new dose until monitoring is stopped
* V7: 12 weeks after starting glargine, the patient presents again for placement of the CGM device (start of monitoring). The patient will also do a glycemic cycle at the same time and communicate it to his ARC. A laboratory assessment (including glycated hemoglobin) will be requested.
* V8: 12 weeks + 7 days stop CGM monitoring (collection of holter results under glargine) and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 and <70
* Type 2 diabetic patients, with a duration of NPH between 5 and 10 years.
* Patients treated with a double dose of NPH insulin with a stable dose of insulin and a stable dose of ADO (oral antidiabetic drugs) for at least 2 months prior to the start of the study.
* An HbA1c level between 7% and 10%
* Ability to use a continuous glucose monitoring (CGM) system and cycle blood glucose with the meter.
* Written informed consent obtained prior to participation in the study.

Exclusion Criteria:

* Pregnant and breastfeeding women
* Patients with active proliferative and/or complicated diabetic retinopathy, treated by photocoagulation or surgically, within 6 months prior to study entry or any other rapidly progressing unstable retinopathy that may require photocoagulation or surgery during the study (plan to perform fundus prior to inclusion).
* History of insulin glargine hypersensitivity
* Treatment with systemic, neuroleptic, immunosuppressive and antiretroviral corticosteroids within 3 months prior to study entry and during the study and other treatments, which may significantly affect blood glucose.
* Severe renal impairment at baseline defined by a < 30ml/min.
* Patients on sulfonylurea drugs or glinides or on more than three oral antidiabetic drugs (ODAs)
* Patients on rapid insulin.
* Patients Enrolled in Other Clinical Studies
* Patients who refuse to sign consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
glycaemic variability on insulin glargine (after 12 weeks of use) versus NPH insulin (baseline) | 4 months
  compare glycaemic variability on insulin glargine (after 12 weeks of use) versus NPH insulin (baseline) using the CGM device generating the area under the curve in the range, above the range, below the range in type 2 diabetic patients treated with NPH basal insulin alone or in combination with oral antidiabetic drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Rekik, Professor, Principal Investigator — STEDIAM
Locations (1):
- Hedi Chaker Hospital, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cohen MP, Shea E, Chen S, Shearman CW. Glycated albumin increases oxidative stress, activates NF-kappa B and extracellular signal-regulated kinase (ERK), and stimulates ERK-dependent transforming growth factor-beta 1 production in macrophage RAW cells. J Lab Clin Med. 2003 Apr;141(4):242-9. doi: 10.1067/mlc.2003.27. PMID 12677169
- [Result] Danielsson P, Truedsson L, Eriksson KF, Norgren L. Inflammatory markers and IL-6 polymorphism in peripheral arterial disease with and without diabetes mellitus. Vasc Med. 2005 Aug;10(3):191-8. doi: 10.1191/1358863x05vm617oa. PMID 16235772
- [Result] Hirsch IB, Brownlee M. Should minimal blood glucose variability become the gold standard of glycemic control? J Diabetes Complications. 2005 May-Jun;19(3):178-81. doi: 10.1016/j.jdiacomp.2004.10.001. PMID 15866065